CLINICAL TRIAL: NCT05211258
Title: A Novel Portable Upper Gastrointestinal Endoscopy System Applied in Remote Populations: A Pilot Study
Brief Title: A Novel Portable Upper Gastrointestinal Endoscopy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: portable-endo
Record Dates: First submitted 2021-12-27; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Digestive System Disease; Diagnoses Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a novel portable upper gastrointestinal endoscopy system (Experimental)
  Interventions: Device: a novel portable upper gastrointestinal endoscopy system

INTERVENTIONS:
Device: a novel portable upper gastrointestinal endoscopy system — Patients arrived at the hospital in the morning after an overnight fast (>6 hours). The patients took oral dyclonine glue 15 mins before their examination. The doctors prepared the portable endoscopy system so that it was in working status and the disposable sheathed system was placed on the endoscope optical probe.

SUMMARY:
The application of conventional endoscopy in remote and outdoor areas lacking facilities remains challenges. Thus, the investigators developed a novel portable upper gastrointestinal endoscopy system that has the same functions as conventional endoscopy. A total of 24 participants from a medical unit on a remote island in China underwent endoscopy with the portable system between March and June 2021. The portable system packed into a suitcase is 68 × 42 × 32 cm in size, weighing less than 35 kg, and comprises a disposable sheathed system.

DETAILED DESCRIPTION:
The application of conventional endoscopy in remote and outdoor areas lacking facilities remains challenges. Thus, the investigators developed a novel portable upper gastrointestinal endoscopy system that has the same functions as conventional endoscopy. A total of 24 participants from a medical unit on a remote island in China underwent endoscopy with the portable system between March and June 2021. The portable system packed into a suitcase is 68 × 42 × 32 cm in size, weighing less than 35 kg, and comprises a disposable sheathed system. The examination time and any malfunctions in the portable endoscopy system during the examination were recorded. After the examination was finished, the disposable sheathed system was removed, and a pressure leak test was performed to check the seal of the system. The patients were followed up within three days to confirm any adverse events such as nausea, vomiting, throat discomfort, bleeding, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopy examination with the portable system were aged from 18-70 years and presented with upper abdominal complaints.

Exclusion Criteria:

* The exclusion criteria were the same as the contraindications for conventional upper GI endoscopy and included latex allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The examination time | 24 hours
  duration from the time the endoscope was inserted into the patient's mouth to the time it was withdrawn.

SECONDARY OUTCOMES:
adverse events | one week
  nausea, vomiting, throat discomfort, bleeding, etc
number of malfunctions of portable endoscopy system | 24 hours
  hydropower and gas failure, image display failure, disposable sheathed system damage, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided